CLINICAL TRIAL: NCT00778908
Title: Late-Course Accelerated Hyperfractionated IMRT Versus Conventionally Fractionated IMRT in the Treatment of Locoregionally Advanced Nasopharyngeal Carcinoma: A Prospective Randomized Clinical Trial
Brief Title: Late-Course Accelerated Hyperfractionated IMRT for Locoregionally Advanced Nasopharyngeal Carcinoma
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Guangxi Medical University (Other)
Collaborators: People's Hospital of Guangxi Zhuang Autonomous Region (Other); Guangxi Sci-Tech Office (Unknown)
Responsible Party: Principal Investigator, Heming Lu, Associate Professor, People's Hospital of Guangxi Zhuang Autonomous Region
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GUIKEGONG-0816004-40
Record Dates: First submitted 2008-10-22; First posted 2008-10-24 (Estimated); Last update posted 2012-08-21 (Estimated); Status verified 2012-08

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Nasopharyngeal carcinoma; Locally advanced disease; Intensity-modulated radiation therapy; Accelerated hyperfractionation; Concomitant boost radiation therapy; Concurrent chemotherapy
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Late-course accelerated hyperfractionated IMRT with concomitant cisplatin chemotherapy
  Interventions: Radiation: Late-course accelerated hyperfractionated IMRT; Drug: Concomitant cisplatin chemotherapy
- B (Other): Conventionally fractionated IMRT with concomitant cisplatin chemotherapy
  Interventions: Drug: Concomitant cisplatin chemotherapy; Radiation: Conventionally fractionated IMRT

INTERVENTIONS:
Radiation: Late-course accelerated hyperfractionated IMRT — 1. IMRT target definition: PTV1=Gloss tumor PTV; PTV2=High risk area containing subclinical disease; PTV3=Low risk area containing subclinical disease
  2. IMRT delivery scheduling: (1) Six-week treatment: PTV1=60Gy/30fractions, PTV2=57Gy/30fractions,PTV3=54Gy/30fractions.(2) Concomitant boost to PTV1 as a second daily treatment for the last 10 treatments of the Six-week treatment: PTV1=12Gy/10fractions.(3) PTV3 will be treated with conventional radiotherapy technique separately.
  Arms: A
Drug: Concomitant cisplatin chemotherapy — cisplatin:40mg/m2 weekly infusion for 6 weeks
Radiation: Conventionally fractionated IMRT — IMRT target definition: PTV1=Gloss tumor PTV; PTV2=High risk area containing subclinical disease; PTV3=Low risk area containing subclinical disease IMRT delivery scheduling: (1) Seven-week treatment: PTV1=70Gy/35fractions, PTV2=63Gy/35fractions,PTV3=55.8Gy/31fractions.(2) PTV3 will be treated with conventional radiotherapy technique separately.
  Arms: B

SUMMARY:
Based on the radiobiological findings that accelerated tumor repopulation in nasopharyngeal carcinoma occurs in the late-course of radiation therapy, the investigators hypothesize that intensity-modulated radiation therapy(IMRT) with concomitant boost schedule by increasing daily dose starting at the fifth week after initiation of IMRT might improve tumor control and decrease treatment toxicities for locoregionally advanced nasopharyngeal carcinoma. The study is designed to test if late-course accelerated hyperfractionated IMRT can improve the outcomes as compared with conventionally fractionated IMRT in newly diagnosed patients with locoregionally advanced nasopharyngeal carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven non-keratinizing or undifferentiated type nasopharyngeal carcinoma for primary treatment with curative intent
* According to AJCC 2002 Staging System, clinical stage must be Ⅱb-Ⅳb
* Age between 18-70
* Karnofsky performance status ≥70
* WBC ≥4,000/mm3, PLT ≥ 100,000/mm3,serum creatinine ≤ 1.6 mg/dl
* Without radiotherapy or chemotherapy
* Signed study-specific consent form prior to study entry

Exclusion Criteria:

* Patients with distant metastasis
* Pregnant or lactating women
* The presence of uncontrolled life-threatening illness
* Patients who received radiotherapy or chemotherapy previously

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2008-01; Primary Completion 2011-01 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Local/regional control rate, Acute and late toxicities | 2-Yr

SECONDARY OUTCOMES:
Overall survival rate | 5-Yr

CONTACTS AND LOCATIONS:
Overall Officials: Heming Lu, MD, Study Chair — Department of Radiation Oncology, People's Hospital of Guangxi Zhuang Autonomous Region
Locations (1):
- People's Hospital of Guangxi Zhuang Autonomous Region, Nanning, Guangxi, China

REFERENCES:
- See also: Guangxi Sci-Tech Office — http://www.gxsti.net.cn/GXSAT/Default.shtml
- See also: Guangxi Medical University — http://www.gxmu.edu.cn/